CLINICAL TRIAL: NCT04927533
Title: Improving Cognitive and Emotional Processing in Older (Psychiatric) Patients: the Transdiagnostic Effectiveness of the Ronnie Gardiner Method (RGM).
Brief Title: The Ronnie Gardiner Method Effectiveness Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Psychiatric Clinic of Alexianen Zorggroep Tienen (Unknown)
Responsible Party: Principal Investigator, Xenia Brancart, PhD student, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: B.U.N. 1432021000379
Record Dates: First submitted 2021-06-02; First posted 2021-06-16 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Psychiatric Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Older adults with psychiatric problems (Experimental): The target group is a group of older adults with psychiatric problems (≥60 years old) admitted to a residential psychogeriatric department of the Psychiatric Clinic of the Alexians Care Group Tienen. The following exclusion criteria apply: a score of less than 21 on the MMSE (excluding dementia or other moderate to severe cognitive disorders), a mother tongue other than Dutch and having undergone surgery and/or chemotherapy in the last 3 months.
  Interventions: Other: Ronnie Gardiner Method

INTERVENTIONS:
Other: Ronnie Gardiner Method — The Ronnie Gardiner Method (RGM), developed in 1993 by Swedish jazz drummer Ronnie Gardiner, is a promising multimodal, music-based intervention with potential to stimulate and improve several cognitive functions, motor skills, reading and speech skills and social interaction. RGM participants are required to follow (what is known as) "choreoscores". This is a visual representation of the sequence of movements using four unique symbols. Each symbol represents a body half via color (red = left side, blue = right side) and the use of a body part via shape (the symbols resemble hands or feet). In addition, each movement has a specific name, based on drum sounds, which must be pronounced simultaneously. The exercises are guided by trained 'RGM-practitioners'. The course and difficulty of the session can be adapted in different ways by the RGM Practitioner, according to the capabilities of the participants.
  Other Names: RGM (abbreviation)

SUMMARY:
The investigators want to investigate the feasibility and transdiagnostic effectiveness of the Ronnie Gardiner Method (RGM) in a sample of Flemish psychogeriatric residential patients (≥60 years old) admitted to the Psychiatric Clinic of Alexianen Zorggroep Tienen. No control group will be used in this study, as every patient in the clinic is entitled to receive treatment. The investigators expect to observe significant improvements in the core executive functions (core EFs) by RGM participation. The investigators expect that the more sessions participants follow, the larger the effects will be. Given the strong connection between executive functions and emotion regulation, the investigators anticipate that strengthening the core EFs will in turn contribute to better emotion regulation. More specifically, the mediating role of core EFs in the relationship between the number of RGM sessions attended and improvement in emotion regulation is investigated. Given RGMs previously reported effects on quality of life, the investigators also expect to observe improved well-being. Additionally, the investigators want to examine to what extent positive experiences with RGM and temperament based personality types influence the effectiveness of the RGM training.

The RGM training will be organised twice a week for a period of 12 weeks. The training sessions will be provided by trained RGM-practitioners in the Psychiatric Clinic of the Alexianen Zorggroep Tienen. Each session will last at least 45 minutes. Core EFs, emotion regulation and well-being are evaluated pre-, mid- and post-RGM (at 6-week intervals) using a number of relevant instruments (i.e. questionnaires and neuropsychological tests). At baseline, the information and consent forms will be delivered to the patient and exclusion criteria will be checked using the MMSE and the patient file. Experiences with RGM training will be evaluated midway and post-intervention by means of a brief questionnaire developed by the research team. Personality type questionnaires (The Behavioural Inhibition System (BIS)/Behavioural Activation System (BAS) scales and the Effortful Control (EC) scale), which allow us to study whether a particular temperament based personality type is predictive of RGMs success, are routinely administered in the psychiatric clinic upon admission.

ELIGIBILITY:
Inclusion Criteria:

* Psychogeriatric inpatients aged 60+

Exclusion Criteria:

* Checking for moderate to severe cognitive impairments (exclusion criterion) using the Mini-Mental State Examination (MMSE; Folstein, Folstein, & McHugh, 1975; Dutch version: Kok and Verhey, 2002), following exclusion criterion applies: a score of less than 21 on the MMSE (excluding dementia or other moderate to severe cognitive impairment)
* Not fluent in Dutch
* Having undergone surgery and/or chemotherapy in the last three months.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in Emotion Regulation using the Cognitive Emotion Regulation Questionnaire (CERQ; Garnefski, Kraaij & Spinhoven, 2002) | before the start of RGM-training, after 6 weeks of RGM-training and after 12 weeks of RGM-training
  The CERQ was originally developed in Dutch. This self-report questionnaire has 36 items that evaluate the frequency of the use of emotion regulation strategies. The items are divided proportionally among nine emotion regulation strategies based on theory and empirical research: blaming yourself, blaming others, accepting, rumination, relating, catastrophising, focusing on other positive things, focusing on planning and positively reinterpreting. The items are answered on a Likert five-point scale ranging from almost never (1) to almost always (5) (Kraaij & Garnefski, 2006; Garnefski & Kraaij, 2006; Garnefski & Kraaij, 2007; Nowlan et al., 2015). Variations in the total scores of the nine subscales of the CERQ will be examined.
Change in Core EFs (i.e. motor/response inhibition, cognitive flexibility and working memory) using four subtests of the Cambridge Neuropsychological Test Automated Battery (CANTAB® [Cognitive assessment software]). | before the start of RGM-training, after 6 weeks of RGM-training and after 12 weeks of RGM-training
  The four subtests are: (1)Intra-Extra Dimensional Set Shift (Cognitive Flexibility), (2) Spatial Span, (3) Spatial Working Memory and (4) Stop-Signal Task (Inhibition).
  For the subtest Intra-Extra Dimensional Set Shift (IED), total latency (which is the sum of the response times over all trials) and in addition the total number of errors adjusted (which is the number of incorrect stimulus choices) will be analyzed. Next outcome measure is the Spatial Span Forward Span Length (SSPFSL), which is the longest sequence that the participant can reproduce forward. The Spatial Working Memory Total Errors (SWMTE) is another outcome measure to analyze recall problems. This is a measure of the total number of selections from a box that certainly cannot contain a token. The final outcome measure of the CANTAB is the Stop Signal Task Stop Signal Reaction Time (SSTSSRT), which is the estimated time in which a participant can successfully inhibit their responses 50% of the time.
Change in Core EFs (i.e. cognitive inhibition) using the California Older Adult Stroop Test (COAST) | before the start of RGM-training, after 6 weeks of RGM-training and after 12 weeks of RGM-training
  The COAST is a modified Stroop Color-Word Test (SCWT) that was developed specifically for older adults by Pachana and colleagues (2004). In the COAST, only three, more easily distinguishable colours (red, yellow and green) and a larger font are used to minimise the risk of errors due to colour confusion or reduced visual acuity. In addition, the number of items in the COAST was reduced (to 50 items) to minimise fatigue. For this study, we are mainly interested in the last subtest. In this subtest, colour words are presented in a different ink colour (e.g. the word GREEN with a red ink colour) and the aim is for the participants to name the ink colour and inhibit the reading automaticity. The interference score, total completion time and total error score on the interference task of the COAST will be analyzed in this study.
  Thus, both response/motor inhibition (using the CANTAB Stop-Signal Task) and cognitive inhibition (using the COAST) are studied.
Monitor mental well-being using the Dutch version of the 14-item Warwick-Edingburgh Mental Well-Being Scale (WEMWBS) | before the start of RGM-training, after 6 weeks of RGM-training and after 12 weeks of RGM-training
  This questionnaire includes 14 (positively worded) items that question mental well-being (Taggart & Stewart-Brown, 2015; Tennant et al., 2007). The questionnaire is suitable for individuals as young as 13 years old (Taggart & Stewart-Brown, 2015). Participants are required to answer the items on a five-point scale, ranging from never (1) to always (5), according to their psychological functioning over the past two weeks. The sensitivity to change of the WEMWBS has been well validated (Taggart & Stewart-Brown, 2015). This is important in intervention studies where pre- and post-scores are compared, which is also the aim in the current study. The research duo Taggart and Stewart-Brown (2015) compared different instruments of mental well-being and concluded that the WEMWBS is preferred (over the WHO-5) in intervention studies.
  The total score will be analyzed for this study. The higher the total score, the higher the level of mental well-being (Tennant et al., 2007).

SECONDARY OUTCOMES:
Defining the temperament based personality type using the Behavioural Inhibition System (BIS)/Behavioural Activation System (BAS) scale | routinely administrated in the psychiatric clinic upon admission
  The BIS/BAS scale is a Dutch personality questionnaire that assesses fear-related avoidance behavior (BIS scale) and reward-related approach behavior (BAS scale) (Gray, 1970). The 24 items can be subdivided into four scales, three of which are related to the BAS scale (i.e. fun seeking, drive en reward responsiveness) and lastly the BIS scale (Franken et al., 2005).
  The BIS and BAS total scores will be used to determine membership to a particular personality type.
Experiences with RGM-training | after 6 weeks of RGM-training and after 12 weeks of RGM-training
  In order to investigate the contribution of positive experiences to the effectiveness of RGM, the research team has developed a short questionnaire. This questionnaire includes three questions that directly and indirectly question the experiences in RGM. The three questions are: "To what extent do you find the RGM training enjoyable?", "To what extent would you recommend the RGM training to your fellow patients?" and "To what extent would you participate in the RGM training again?". Participants should answer the questions on a ten-point scale ranging from "not at all" (1) to "very much" (10). The higher the total score (outcome measure), the higher the positive experience of the RGM training.
Defining the temperament based personality type using the Effortful Control (EC) scale | routinely administrated in the psychiatric clinic upon admission
  The 19-item Effortful Control Scale (ECS; Evans & Rothbart, 2007; Dutch version, Hartman & Rothbart, 2001) is a scale of the Adult Temperament Questionnaire (ATQ) that questions the extent to which an individual can direct his or her attention (i.e. attention control), can activate a response (i.e. activation control) and the ability to inhibit inappropriate behavior (i.e. inhibitory control). The three subscales of the ECS reflect the aforementioned concepts.
  The EC total score will be used to determine membership to a particular personality type.

CONTACTS AND LOCATIONS:
Overall Officials: Xenia Brancart, Principal Investigator — Vrije Universiteit Brussel - Ghent University; Gina Rossi, Prof. Dr., Principal Investigator — Vrije Universiteit Brussel; Eva Dierckx, Prof. Dr., Principal Investigator — Vrije Universiteit Brussel - Alexianen Zorggroep Tienen; Rudi De Raedt, Prof. Dr., Principal Investigator — University Ghent
Locations (1):
- Alexianen Zorggroep Tienen, Tienen, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pohl P, Dizdar N, Hallert E. The Ronnie Gardiner Rhythm and Music Method - a feasibility study in Parkinson's disease. Disabil Rehabil. 2013;35(26):2197-204. doi: 10.3109/09638288.2013.774060. Epub 2013 Mar 12. PMID 23480646
- [Background] Thornberg K, Josephsson S, Lindquist I. Experiences of participation in rhythm and movement therapy after stroke. Disabil Rehabil. 2014;36(22):1869-74. doi: 10.3109/09638288.2013.876107. Epub 2014 Jan 9. PMID 24400709
- [Background] Bunketorp-Kall L, Lundgren-Nilsson A, Samuelsson H, Pekny T, Blomve K, Pekna M, Pekny M, Blomstrand C, Nilsson M. Long-Term Improvements After Multimodal Rehabilitation in Late Phase After Stroke: A Randomized Controlled Trial. Stroke. 2017 Jul;48(7):1916-1924. doi: 10.1161/STROKEAHA.116.016433. Epub 2017 Jun 15. PMID 28619985